CLINICAL TRIAL: NCT06336603
Title: The Combination Use of Winlevi and Adapalene 0.3% Gel in Real Life Acne Treatment
Brief Title: A Study Assessing the Efficacy of Combined Use of Clascoterone 1% Cream and Adapalene 0.3% for the Treatment of Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIN2022
Record Dates: First submitted 2024-03-11; First posted 2024-03-29 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone; Adapalene; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Winlevi (clascoterone) 1% & Adapalene 0.3% gel (Experimental): Combined use of Winlevi twice daily and Adapalene once daily
  Interventions: Drug: Winlevi (clascoterone) 1% & Adapalene 0.3% gel

INTERVENTIONS:
Drug: Winlevi (clascoterone) 1% & Adapalene 0.3% gel — Participants will use Winlevi (clascoterone) 1% twice daily (BID) and Adapalene 0.3% once daily (QD)

SUMMARY:
Winlevi is the first topical anti androgen and sebum inhibitor approved for acne vulgaris. There is no study assessing Winlevi in combination treatment for acne .Therefore this study assesses Winlevi with Adapalene 0.3% gel in combination to emulate real life practice.

ELIGIBILITY:
Inclusion Criteria:

i. Outpatient, male or female subjects of any race, and at least 12 years of age or older.

* Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline (test must have a sensitivity of at least 25mIU/ml for human chorionic gonadotropin) and practice a reliable method of contraception throughout the study:
* A female is considered of childbearing potential unless she is:

  1. postmenopausal for at least 12 months prior to study drug administration;
  2. without a uterus and/or both ovaries; or
  3. Has been surgically sterile for at least 6 months prior to study drug administration.
* Reliable methods of contraception are:

  1. Hormonal methods or intrauterine device in use > 90 days prior to study drug administration;
  2. Barrier methods plus spermicide in use at least 14 days prior to study drug administration; or
  3. Vasectomized partner (vasectomy must be performed 3 months prior to first study drug administration or in the alternative a zero sperm count will suffice).
* Exception: Female subjects of childbearing potential who are not sexually active will not be required to practice a reliable method of contraception. These subjects may be enrolled at the Investigator's discretion if they are counseled to remain sexually inactive during the study and understand the possible risks in getting pregnant during the study.

ii. Facial acne IGA score of 3 or 4.

iii. Able to understand the requirements of the study and sign Informed Consent/HIPAA Authorization forms. Subjects under the legal age of consent in the state where the study is conducted must also have the written, informed consent of a parent or legal guardian.

Exclusion Criteria:

i. Female subjects who are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.

ii. Allergy or sensitivity to any component of the test medications (Section 5.2).

iii. Subjects who have not complied with the proper wash-out periods for prohibited medications (Supplement I).

iv. Medical condition that, in the opinion of the Investigator, contraindicates the subject's participation in the clinical study.

v. Skin disease/disorder that might interfere with the diagnosis or evaluation of acne vulgaris vi. Evidence of recent alcohol or drug abuse. vii. History of poor cooperation, non-compliance with medical treatment, or unreliability.

viii. Exposure to an investigational drug study within 30 days of the Baseline Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Sciences, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Started | 20
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black | 4
  Asian | 4
  Hispanic | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study is the Percent of Patients Who Achieve Clear or Almost Clear on IGA at Week 16.
Description: The investigator will evaluate global acne severity using the Investigator Global Assessment scale, which ranges from 0 to 5, where 0 represents clear skin and 5 represents very severe acne
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants | 65

2. Secondary Outcome: Percent of Total Lesion Reduction at Week 16 Compared to Baseline
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
Percentage change | 87.3 (11.4)
Statistical Analysis 1: Comparison: Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel; Test type: Superiority; p < .001, Wilcoxon signed rank test

3. Secondary Outcome: Percent of Inflammatory Lesion Reduction at Week 16 Compared to Baseline
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage change | 90.5 (10.1)
Statistical Analysis 1: Comparison: Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel; Test type: Superiority; p < .001, Wilcoxon signed rank test

4. Secondary Outcome: Percent of Non-inflammatory Lesion Reduction at Week 16 Compared to Baseline
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage change | 84.8 (13.5)
Statistical Analysis 1: Comparison: Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel; Test type: Superiority; p < .001, Wilcoxon signed rank test

5. Secondary Outcome: Tolerability Measures of Erythema Based on 5-point Severity Scale
Description: The score in the scale ranges from 0-4. Lower score represents absence of erythema and higher score represents severe condition.
  The information presented represents the "Percentage of participant" with "Absent or Trace" erythema at weeks 4,8,12, 16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 76
  Week 4 | 88
  Week 8 | 100
  Week 12 | 100
  Week 16 | 94
  Week 20 | 100

6. Secondary Outcome: Tolerability Measures of Dryness Based on 5-point Severity Scale
Description: The score in the scale ranges from 0-4. Lower score represents absence of dryness and higher score represents severe condition.
  The information presented represents the "Percentage of participant" with "Absent or Trace" Dryness at weeks 4,8,12, 16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 100
  Week 4 | 100
  Week 8 | 100
  Week 12 | 100
  Week 16 | 100
  Week 20 | 100

7. Secondary Outcome: Tolerability Measures of Peeling Based on 5-point Severity Scale
Description: The score in the scale ranges from 0-4. Score 0 represents absence of peeling and Score 4 represents 'Extensive peeling'.
  The information presented represents the "Percentage of participant" with "Absent or Trace" peeling at weeks 4,8,12,16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 100
  Week 4 | 100
  Week 8 | 100
  Week 12 | 100
  Week 16 | 100
  Week 20 | 100

8. Secondary Outcome: Assessment of Skin Oiliness Based on 5-point Severity Scale
Description: The score in the scale ranges from 0-4. Score 0 represents absence of Oiliness and Score 4 represents severe condition.
  The information presented represents the "Percentage of participant" with "Absent or Trace" oiliness at weeks 4,8,12,16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 76
  Week 4 | 82
  Week 8 | 94
  Week 12 | 94
  Week 16 | 94
  Week 20 | 94

9. Secondary Outcome: Tolerability Measures of Burning/Stinging Based on 6-point Severity Scale
Description: The score in the scale ranges from 0-5. Lower score represents absence of discomfort and higher score represents severe condition.
  The information presented represents the "Percentage of participant" with "Absent or Trace" burning/stinging at weeks 4,8,12,16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 100
  Week 4 | 100
  Week 8 | 94
  Week 12 | 94
  Week 16 | 100
  Week 20 | 100

10. Secondary Outcome: Tolerability Measures of Pruritus Based on 6-point Severity Scale
Description: The score in the scale ranges from 0-5. Lower score represents absence of discomfort and higher score represents severe condition.
  The information presented represents the "Percentage of participant" with "Absent or Trace" pruritus at weeks 4,8,12,16 and 20
Time Frame: Week 4,8,12,16, 20
Measure: Number; unit: percentage of participants
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
Number analyzed (Participants) | 17
percentage of participants
  Baseline | 94
  Week 4 | 88
  Week 8 | 88
  Week 12 | 94
  Week 16 | 94
  Week 20 | 100

ADVERSE EVENTS:
Time Frame: 20 Weeks
Arm/Group | Winlevi (Clascoterone) 1% & Adapalene 0.3% Gel
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT06336603/Prot_SAP_000.pdf